CLINICAL TRIAL: NCT04473833
Title: Transvaginal Ultrasonography as a Screening Method for Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John R van Nagell (Other)
Responsible Party: Sponsor-Investigator, John R van Nagell, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MCC-88-GYN-13
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer
Keywords: serial; transvaginal ultrasonography
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants in the Kentucky Ovarian Cancer Screening Program (Experimental): Participants from the Kentucky Ovarian Cancer Screening Program who choose to participate in this trial will undergo further serial transvaginal ultrasonography (TVS) screening.
  Interventions: Procedure: Serial Transvaginal Ultrasonography

INTERVENTIONS:
Procedure: Serial Transvaginal Ultrasonography — Participants will undergo transvaginal ultrasonography (TVS) to detect ovarian cancer as part of the Kentucky Ovarian Cancer Screening Program. Those with normal findings will repeat the TVS in one year. Those with abnormal results will repeat the screening in 4-6 weeks.

SUMMARY:
This is a large, prospective, single-arm cohort study of transvaginal ultrasonographic screening for ovarian cancer in intermediate to high-risk women from Kentucky. Detection of ovarian malignancy often occurs subsequent to the initial transvaginal sonography (TVS) screen; therefore, it is important to offer continued screening to study participants based on our published algorithm. Screening will be available to participants for as long as they elect to receive it. The primary study endpoints are to determine if prospective serial transvaginal ultrasonography can decrease the false-positive (FP) percentage and improve the positive predictive value (PPV) as suggested by retrospective analysis without compromising the detection of true positives or promote the occurrence of false negatives.

DETAILED DESCRIPTION:
Women from every Kentucky county participate in the Kentucky Ovarian Cancer Screening Program. Screening sites include: Maysville, Prestonsburg, Greenup, Elizabethtown, Somerset, Paducah and Lexington. Offsite participants account for 14% of the screening population with 86% being screened in Lexington. The long-term survival (20 year) of women with screen-detected ovarian cancers is twice that of unscreened women (65% vs 32%). Separation of cases into Type 1 and Type 2 ovarian cancer shows that screening improves the survival of both Type 1 and Type 2 ovarian cancers. Type 1 ovarian carcinomas for the screened and unscreened populations were defined based on these WHO criteria: mucinous carcinomas all grade, clear cell carcinomas all grades, endometrioid carcinomas grades 1 & 2, serous carcinomas grades 1 & 2, and malignant Brenner's tumors all grades. Type 2 ovarian carcinomas for the screened and unscreened populations were defined based on these criteria: undifferentiated carcinomas, endometrioid carcinomas grade 3, serous carcinomas grade 3, and carcinosarcomas.

While long-term 20-year survival of women with Type 1 ovarian cancers detected by screening was significantly better than for unscreened women (81% v 46%, respectively), the survival benefit was even more pronounced for Type 2 ovarian cancers detected by screening of Kentucky women compared to unscreened Kentucky women (55.7% vs. 0.3%, respectively) or unscreened women at UK Hospital (12%). Screen-detected cases of Type 2 invasive ovarian cancers had better survival than unscreened cases when those detected had early- or late-stage disease. However, better survival was achieved when Type 2 ovarian cancers were detected at an early (72%) compared to late-stage (46%). Our data support the effectiveness of the screening protocol at the University of Kentucky, and subsequent treatment in accordance with National Comprehensive Cancer Network guidelines.

The significance of these findings is that our approach has resulted in the detection of both early-stage Type 1 and Type 2 ovarian cancers and these cases have had improved survival when compared to that of unscreened cases, indicating that the screen-detected cases are associated with a potential survival advantage even for aggressive ovarian carcinomas.

The primary objective of this study is to prospectively evaluate the false positive (FP) percentage generated by the ovarian screening algorithm and determine whether serial transvaginal ultrasonography can lower the FP percentage as demonstrated in the retrospective analysis. The aim of serial ultrasonography is to decrease FP percentage to 0.32% (positive predictive value of 24%) without adversely impacting the results for true positives and false negatives. on a "per woman screened basis" since this corresponds to a minimally acceptable positive predictive value of 24% or higher. This assumes an average of three screening years for each new woman entering the program.

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 50 years;
* women with a documented family history of ovarian cancer over the age of 24 years;
* women over the age of 24 years with a personal history of breast cancer
* ECOG performance status of 0 to 2.34
* Subjects having undergone prior hysterectomy will be eligible provided that they meet the other requirements for entry into this study and have at least one ovary.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are referred with pelvic symptoms, a known pelvic mass or a history of prior radiation.
* Individuals that cannot safely receive transvaginal ultrasound due to vaginal size, vaginal infections, lack of bowel or bladder control or inability to physically place their body in position to receive transvaginal ultrasound
* Prisoners
* Pregnant women
* Women with a prior history of ovarian cancer
* Exclusions will apply to anyone who presents with factors or issues that prevent them from understanding the screening research procedures or completing the informed consent component or personal information needed for the study

Min Age: 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65000 (Estimated)
Dates: Start 1988-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
False-positive (FP) percentage | approximately 3 years
  Measure the false-positive (FP) rate generated by the ovarian screening algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: John R Van Nagell, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lasher A, Harris LE, Solomon AL, Harbin LM, Raby L, Dietrich CS, Kryscio RJ, van Nagell JR, Pavlik EJ. Variables Associated With Resolution and Persistence of Ovarian Cysts. Obstet Gynecol. 2023 Dec 1;142(6):1293-1301. doi: 10.1097/AOG.0000000000005411. Epub 2023 Oct 12. PMID 38051292